CLINICAL TRIAL: NCT02230033
Title: An Open-Label, Randomized, Parallel-Group Drug-Drug Interaction Study to Assess the Effect of Multiple Doses of Itraconazole or Gemfibrozil on the Pharmacokinetics of a Single Dose of JNJ-56021927 in Healthy Male Subjects
Brief Title: Study to Assess Drug-Drug Interaction Between Itraconazole or Gemfibrozil and JNJ-56021927
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aragon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR105398; 56021927PCR1012 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
Keywords: JNJ-56021927; Itraconazole; Gemfibrozil
MeSH Terms: interventions — Itraconazole; Gemfibrozil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): Single oral dose of JNJ-56021927 240 milligram (mg) capsule will be administered on Day 1.
  Interventions: Drug: JNJ-56021927
- Treatment B (Experimental): Itraconazole 200 mg (2 capsules of 100 mg) will be administered once daily orally from Day 1 until Day 32, along with single oral dose of JNJ-56021927 240 mg capsule on Day 4.
  Interventions: Drug: JNJ-56021927; Drug: Itraconazole
- Treatment C (Experimental): Gemfibrozil 600 mg oral tablet will be administered twice daily from Day 1 until Day 32, along with single oral dose of JNJ-56021927 240 mg capsule on Day 4.
  Interventions: Drug: JNJ-56021927; Drug: Gemfibrozil

INTERVENTIONS:
Drug: JNJ-56021927 — Single oral dose of JNJ-56021927 240 milligram (mg) capsule will be administered on Day 1 or Day 4 in any of the treatment.
Drug: Itraconazole — Itraconazole 200 mg (2 capsules of 100 mg) will be administered once daily orally from Day 1 until Day 32.
  Arms: Treatment B
Drug: Gemfibrozil — Gemfibrozil 600 mg oral tablet will be administered twice daily from Day 1 until Day 32.
  Arms: Treatment C

SUMMARY:
The purpose of this study is to assess the effect of multiple doses of itraconazole or gemfibrozil on the pharmacokinetics (the study of the way a drug enters and leaves the blood and tissues over time) of JNJ-56021927 and its metabolites (JNJ 56142060 and JNJ-56142021) in healthy male participants.

DETAILED DESCRIPTION:
This is a single-dose, single-center, open-label (all people know the identity of the intervention), 3-treatment, randomized (study medication assigned to participants by chance) and parallel-group (a medical research study comparing the response in two or more groups of participants receiving different interventions [treatments]) study. The study consists of Screening Phase (that is, 21 days before study commences on Day 1); open-label treatment Phase and end-of-study or early withdrawal assessment. All participants will be randomly assigned to 1 of 3 treatments, that is, Treatment A (single dose of JNJ-56021927 on Day 1), Treatment B (200 milligram [mg] itraconazole once daily from Day 1 up to Day 32 along with single dose of JNJ-56021927 on Day 4), and Treatment C (600 mg gemfibrozil twice daily from Day 1 up to Day 32 along with single dose of JNJ-56021927 on Day 4). Blood samples will be collected for evaluation of pharmacokinetics at pre-dose and post-dose of study treatment. The maximum duration of participation in the study per participant will be approximately 78 days (Treatment A) or 81 days (Treatment B and C). Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Must agree to use an adequate contraception method as deemed appropriate by the Investigator and specified in protocol, always use a condom during sexual intercourse, and to not donate sperm during the study and for 3 months after receiving the study drug
* Body mass index between 18 and 30 kilogram (kg) per square meter, and body weight not less than 50 kg
* Blood pressure (supine for 5 minutes) between 90 and 140 millimeter of mercury (mm Hg) systolic, and no higher than 90 mm Hg diastolic
* A 12-lead electrocardiogram (ECG) consistent with normal cardiac conduction and function at Screening, including: Pulse rate between 45 and 99 beats per minute (bpm); QTc interval less than or equal to (<=) 450 milliseconds; QRS interval of less than (<) 120 milliseconds; PR interval <220 milliseconds; and morphology consistent with healthy cardiac conduction and function
* Nonsmoker within the previous 2 months (calculated from first dosing)

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the Investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, clinical chemistry or urinalysis at Screening or at admission to the study center as deemed appropriate by the Investigator
* Medical history of gallbladder disease (cholecystitis, cholelithiasis, cholecystectomy)
* Presence of sexual dysfunction or any medical condition that would affect sexual function
* Screening serum testosterone level of < 200 nanogram/deciliter (ng/dL)
* Previous history of photoallergy or phototoxic reaction during treatment with fibrates

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | Up to Day 57 or Day 60
  The Cmax is the maximum observed plasma concentration. Blood samples will be collected up to Day 57 (for Treatment A) or Day 60 (for Treatment B and C).
Time to Reach Maximum Concentration (tmax) | Up to Day 57 or Day 60
  The tmax is time to reach the maximum observed plasma concentration. Blood samples will be collected up to Day 57 (for Treatment A) or Day 60 (for Treatment B and C).
Area Under the Plasma Concentration-Time Curve From Time Zero to 672 Hours (AUC [0-672]) | Up to Day 57 or Day 60
  The AUC (0-672) is the area under the plasma concentration-time curve from time zero to 672 hours. Blood samples will be collected up to Day 57 (for Treatment A) or Day 60 (for Treatment B and C).
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) | Up to Day 57 or Day 60
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time. Blood samples will be collected up to Day 57 (for Treatment A) or Day 60 (for Treatment B and C).
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | Up to Day 57 or Day 60
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z), wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time; C(last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant. Blood samples will be collected up to Day 57 (for Treatment A) or Day 60 (for Treatment B and C).
Percentage of Extrapolated AUC (0-infinity) | Up to Day 57 or Day 60
  The percentage of AUC (0-infinity) that is due to extrapolation from Tlast to infinity (AUC%Extrapolation) is calculated by using the formula AUC_%extrapolation = 100*(AUC [0-infinity] minus (AUC [0-last])/(AUC (0-infinity). Blood samples will be collected up to Day 57 (for Treatment A) or Day 60 (for Treatment B and C).
Elimination Half-Life (t [1/2] Lambda) | Up to Day 57 or Day 60
  Elimination half-life (t [1/2] Lambda) is associated with the terminal slope (lambda [z]) of the semi logarithmic drug concentration-time curve, calculated as 0.693/lambda(z). Blood samples will be collected up to Day 57 (for Treatment A) or Day 60 (for Treatment B and C).
Rate Constant (Lambda[z]) | Up to Day 57 or Day 60
  Lambda(z) is first-order rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve. Blood samples will be collected up to Day 57 (for Treatment A) or Day 60 (for Treatment B and C).
Time to last quantifiable plasma concentration (tlast) | Up to Day 57 or Day 60
  The tlast is the time to last observed quantifiable plasma concentration. Blood samples will be collected up to Day 57 (for Treatment A) or Day 60 (for Treatment B and C).
Total Plasma Clearance (CL/F) of JNJ-56021927 | Up to Day 57 or Day 60
  Total plasma clearance of drug after extravascular administration, uncorrected for absolute bioavailability, calculated as Dose/AUC (0-infinity) (JNJ-56021927 only). Blood samples will be collected up to Day 57 (for Treatment A) or Day 60 (for Treatment B and C).
Metabolite to Parent Drug Ratio for maximum observed plasma concentration (MPR Cmax) | Up to Day 57 or Day 60
  Metabolite to parent drug ratio for maximum observed plasma concentration will be calculated. Blood samples will be collected up to Day 57 (for Treatment A) or Day 60 (for Treatment B and C).
Metabolite to Parent Drug Ratio for AUC (0 to last) (MPR AUC [0-last]) | Up to Day 57 or Day 60
  Metabolite to parent drug ratio for AUC (0 to last) will be calculated. Blood samples will be collected up to Day 57 (for Treatment A) or Day 60 (for Treatment B and C).
Metabolite to Parent Drug Ratio for AUC (0-infinity) (MPR AUC [0-infinity]) | Up to Day 57 or Day 60
  Metabolite to parent drug ratio for AUC (0-infinity) will be calculated. Blood samples will be collected up to Day 57 (for Treatment A) or Day 60 (for Treatment B and C).

SECONDARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs) | Screening up to Day 57 for treatment A or up to Day 60 for treatment B or C or early withdrawal
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to day 57 for treatment A or up to day 60 for treatment B or C, that are absent before treatment or that worsened relative to pretreatment state.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Tempe, Arizona, United States